CLINICAL TRIAL: NCT04127773
Title: Correct Gastric Tube Placement in Very Low Birth Weight Neonates: Comparison of NEX and NEMU Methods
Brief Title: Correct Gastric Tube Placement in Very Low Birth Weight Neonates
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Chiara Baracetti, Registered Nurse, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: GT PLACEMENT IN VLBW
Record Dates: First submitted 2019-07-14; First posted 2019-10-16 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Gastric Tube Placement
Keywords: VLBW - Very Low Birth Weight Infant; Gastric tube; Enteral nutrition; Prematurity; Nursing
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NEX group: oro gastric tube placement using NEX insertion length predictor
  Interventions: Device: oro gastric tube
- NEMU group: oro gastric tube placement using NEMU insertion length predictor
  Interventions: Device: oro gastric tube

INTERVENTIONS:
Device: oro gastric tube — According to clinical need, an orogastric tube will be inserted at birth using the group method in VLBW infants in whom an umbilical catheter has been placed. An X-ray chest will be performed according to routine clinical practice to assess the position of the umbilical catheter. On the same X-ray the position of the gastric tube will be assessed by a radiologist blinded to the method used for orogastric tube placement.

SUMMARY:
Gastric tube (GT) placement is a recurrent procedure in VLBW infants due to feeding impairment correlated with low birth weight.

Correct GT depth is mandatory to ensure an appropriate and safe enteral feeding: X-ray is the gold standard in order to check GT position, but this cannot be routinely performed due to x-ray exposure risk. Feeding a neonate through a misplaced GT is potentially harmful and may increase morbidity, mortality and hospitalization length.

Nurses estimate GT depth through external measurements. This study aims to identify the most appropriate insertion length predictor for orogastric tube placement in VLBW infants by comparing two different methods.

DETAILED DESCRIPTION:
Several methods have been suggested to estimate orogastric tube insertion length, but none of them has been validated in VLBW infants. The most commonly used methods are NEX (Nose-Ear-Xyphoid) and NEMU (Nose-Ear-Mid-Umbilicus) as predictors of nasogastric tube insertion. For the purpose of the present study NEX and NEMU methods were adjusted for orogastric tube placement.

Hence, primary aim of this study is:

To identify the most appropriate insertion length predictor for orogastric tube placement in VLBW infants by comparing NEX and NEMU methods.

Secondary aim is:

- To develop a new mathematical formula, based on the neonate's weight or length, to predict the insertion length of orogastric tube in VLBW infants

ELIGIBILITY:
Inclusion Criteria:

* Birth Weight ≤1500 grams (Very Low Birth Weight Infants)
* Need for both umbilical catheter and gastric tube positioning at birth

Exclusion Criteria:

* Birth Weight >1500 grams
* Congenital respiratory or gastrointestinal tract malformations (from oral cavity to stomach included)
* Critically unstable preterm infants will be excluded according to nurse or physician evaluation

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: VLBW infants
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Gastric tube position | within 24 hours
  Control on X-ray chest of the gastric tube placement by NEX and NEMU methods

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Baracetti, RN, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Mangiagalli Regina Elena, Milano (ITALY)
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Mangiagalli Regina Elena, Milan, Italy

IPD SHARING:
Plan to Share IPD: No